CLINICAL TRIAL: NCT01809860
Title: Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Sirolimus: A Phase 1, Open-Label, Sequential Study in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Sirolimus in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0020
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Subjects; Pharmacokinetics of Isavuconazole; Pharmacokinetics of Sirolimus
Keywords: isavuconazole; sirolimus; BAL8557; Healthy Volunteers
MeSH Terms: interventions — isavuconazole; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- isavuconazole and sirolimus (Experimental): Single dose of sirolimus on Days 1 and 26, isavuconazole 3 times a day (TID) for 2 days (Days 22 to 23) followed by once a day (QD) for 11 days
  Interventions: Drug: isavuconazole; Drug: sirolimus

INTERVENTIONS:
Drug: isavuconazole — Oral
  Other Names: BAL8557
Drug: sirolimus — Oral
  Other Names: Rapamune

SUMMARY:
The purpose of the study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics (PK) of sirolimus after single dose administration.

DETAILED DESCRIPTION:
Subjects will receive a single dose of sirolimus on Day 1 followed by a 21 day wash-out period (time from sirolimus dosing to isavuconazole dosing). On Days 22 and 23, isavuconazole will be dosed three times daily (TID). On Days 24 through 34, isavuconazole will be administered once daily (QD). All subjects will be administered a single dose of sirolimus on Day 26.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 45 kg and has a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* Results for aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be within the normal range
* The female subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years without menses), or using a medically acceptable double barrier method (e.g. spermicide and diaphragm, or spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study; and is not lactating or pregnant as documented by negative pregnancy tests
* The male subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy and agrees to continue using this method from Screening until 3 weeks after the follow-up visit at the end of the study

Exclusion Criteria:

* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* The subject has a history of tuberculosis or exposure to anyone known or suspected to have tuberculosis or any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering study drug to the subject
* The subject has a positive result for hepatitis C antibodies, hepatitis B surface antigen, or QuantiFERON®-TB Gold test or is known to be positive for human immunodeficiency virus (HIV).
* The subject has a known or suspected allergy to any of the components of the trial products including prednisone or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) within 6 months prior to Screening
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to Day -1, or over-the-counter medications within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, or a positive drug and/or alcohol screen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of sirolimus in whole blood: AUCinf | Days 1 and 26 at predose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours postdose
  Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity (AUCinf)
PK of sirolimus in whole blood: AUClast | Days 1 and 26 at predose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours postdose
  AUC from the time of dosing to the last quantifiable concentration (AUClast)
PK of sirolimus in whole blood: Cmax | Days 1 and 26 at predose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours postdose
  Maximum concentration (Cmax)

SECONDARY OUTCOMES:
Composite of PK variables of sirolimus in whole blood: tmax, Vz/F, CL/F, and t 1/2 | Days 1 and 26 at predose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192 and 216 hours postdose
  Time to attain Cmax (tmax), apparent volume of distribution (Vz/F), apparent body clearance after oral dosing (CL/F), and apparent terminal elimination half-life (t1/2)
PK variable of isavuconazole in plasma: Ctrough | Day 24 and Days 28 through 35 predose
  trough concentration (Ctrough)
Composite of PK variables of isavuconazole in plasma: AUCtau, Cmax, and tmax | Day 25, predose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 16 hours postdose; Day 26 predose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24 and 36 hours postdose
  AUC during the time interval between consecutive dosing (AUCtau)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Covance, Dallas, Texas, United States